CLINICAL TRIAL: NCT06251830
Title: Aumentare il Potere Diagnostico Riducendo la Durata Dell'Esame: MR Fingerprinting Soddisfa le Aspettative?
Brief Title: Increasing Diagnosis Rates While Reducing Examination Time: Can MR Fingerprinting Deliver on Its Promise?
Status: Completed | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Mauro Costagli, Researcher, IRCCS Fondazione Stella Maris
Other Study IDs: GR-2016-02361693; GR-2016-02361693 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2024-01-16; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Neurodevelopmental Disorders; Neurodegenerative Diseases; Brain Tumor; Multiple Sclerosis; Epilepsy
MeSH Terms: conditions — Neurodevelopmental Disorders; Neurodegenerative Diseases; Brain Neoplasms; Multiple Sclerosis; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pediatric patients: Pediatric patients referred to the participating imaging centre for a standard MRI procedure.
  Interventions: Diagnostic Test: MRI exam with Magnetic Resonance Fingerprinting
- Adult Patients: Adult patients referred to the participating imaging centre for a standard MRI procedure, with neurological signs and symptoms.
  Interventions: Diagnostic Test: MRI exam with Magnetic Resonance Fingerprinting
- Healthy Controls: Adult healthy controls
  Interventions: Diagnostic Test: MRI exam with Magnetic Resonance Fingerprinting

INTERVENTIONS:
Diagnostic Test: MRI exam with Magnetic Resonance Fingerprinting — Acquisition of MRI data with technique "Magnetic Resonance Fingerprinting"

SUMMARY:
Magnetic Resonance Imaging (MRI) is an excellent method for diagnosis and staging of brain disease. However, lengthy scan times and sensitivity to patient motion limit its efficacy. To address this, a novel method has recently been demonstrated, called MR Fingerprinting (MRF). The investigators' improved implementation of MRF, featuring fully-quantitative data and a reduced sensitivity to patient motion, can be used to acquire an anatomical exam in less than five minutes at a standard resolution. The potential for wide applicability of this technique, combined with an implied reduction in complexity and cost of MRI exams, has generated wide interest. However, published studies have been limited to demonstrations in healthy volunteers, and the effectiveness of MRF in the clinical practice has not yet been proven. Here, the investigators aim to assess the efficacy of MRF in performing diagnostic exams avoiding sedation in children and for increasing diagnosis rates in challenging adult patients.

DETAILED DESCRIPTION:
Due to its unrivalled diagnostic and prognostic capabilities, as well as the absence of harmful effects from ionizing radiation, MRI is often the radiological method of choice in children. However, radiology units have to face the inability to produce motion-free images especially in young children, even more so in those affected by neurological or neuropsychiatric disorders. These children are often incapable of completely following verbal instructions and cannot remain still in the scanner for a full exam. To avoid uncontrolled motion and the anxiety derived from long examinations, the majority of young children are sedated. However, sedation represents an extra procedure, carrying its own possible adverse effects, procedural complications as well as additional costs. Producing diagnostic, artefact-free images in a short time in children without sedation is thus an unmet need. The investigators' first hypothesis is that MR Fingerprinting can be used in a number of cases to perform a fast and diagnostic exam in children without using sedation.

The advantages of a fast, motion-resistant quantitative scan are not limited to paediatrics but could see wide application.

Disorders of movement such as tremor-dominant Parkinson's disease and severe cognitive impairments such as Alzheimer's disease represent a big challenge when referred to MRI. Although MRI is not a major player in diagnosing such diseases, these patients often require an exam in order to exclude other pathologies with similar clinical manifestations and to diagnose or follow-up other concomitant conditions. Patients with expansive intracranial lesions or requiring frequent follow-up, like those affected by inflammatory disease of the central nervous system, need to undergo long and demanding procedures, and they can eventually get into significant distress. The image quality of standard MRI with these challenging patient groups is often poor, as they cannot lay still or are unable to follow instructions. The investigators' second hypothesis is that MRF can be used to increase diagnosis rates of exams in difficult adult populations, reducing the time spent in the scanner and thus reducing wasted procedures and cost, and increasing patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* ability of understanding and speaking Italian;
* patients referred to the participating imaging centres for a standard MRI procedure;
* adult healthy controls.

For adult patients: inclusion criteria will comprise movement disorders, severe cognitive impairment, expansive intracranial lesions and inflammatory diseases of the central nervous system.

Exclusion Criteria:

* contraindications to the MRI exam

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric patients referred to the participating imaging centre for a standard MRI procedure.
  Adult patients referred to the participating imaging centre for a standard MRI procedure, with neurological signs and symptoms.
  Adult healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 610 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
MRF diagnostic power | "Day 1" - Single time point (MRI examination)
  To evaluate diagnosis rates with MRF in pediatric patients and challenging adult populations

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - IRCCS Stella Maris, Pisa

IPD SHARING:
Plan to Share IPD: No